CLINICAL TRIAL: NCT02063594
Title: Phase 1 Single Dose, Double-blind, Dose-escalation, Safety, Tolerability and Pharmacokinetic Study of NCTX (PEGylated Liposomal Iodixanol Injection) in Healthy Volunteers
Brief Title: Single Dose Safety, Tolerability and Pharmacokinetic Study of NCTX in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Marval Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: MARV2013-CP-001
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers
Keywords: Iodixanol; Iodinated Contrast; Liposome; Computed Tomography; X-ray Imaging; Blood pool agent; Biomarker

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline Placebo (Placebo Comparator): 2 of 8 subjects in each dose cohort will receive normal saline as a single intravenous infusion
  Interventions: Drug: Saline Placebo
- NCTX (Experimental): 6 of 8 subjects in each dose cohort will receive NCTX (PEGylated Liposomal Iodixanol Injection) as a single intravenous infusion
  Interventions: Drug: NCTX (PEGylated Liposomal Iodixanol Injection)

INTERVENTIONS:
Drug: NCTX (PEGylated Liposomal Iodixanol Injection) — Single dose of NCTX (PEGylated Liposomal Iodixanol Injection) administered at escalating doses from 9 mg I/kg up to 110 mg I/kg
  Other Names: NCTX
  Arms: NCTX
Drug: Saline Placebo — Single dose of 0.9% Sodium Chloride Injection, USP administered similarly and at an equivalent dose volume as the active drug
  Arms: Saline Placebo

SUMMARY:
This is a randomized, double-blind, single dose, dose-escalation study to evaluate the safety, tolerability, and pharmacokinetics of NCTX (PEGylated Liposomal Iodixanol Injection) administered intravenously to healthy volunteers. In addition, computed tomography (CT) scans will be acquired to measure radiographic density in regions of interest (ROI) at times from 3-5 hours and up to 72 hours following NCTX administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonsmoking men and women 18 to 55 years of age
* Body Mass Index (BMI) between 18.5 and 30.0 kg/m2
* Serum creatinine within normal range and calculated creatinine clearance of 80 mL/min/1.73 m2 or greater

Exclusion Criteria:

* Concurrent enrollment in another clinical trial or treatment with any investigational products or therapies within 30 days prior to dosing
* History of infusion reactions to liposomes, nanoparticles, monoclonal antibodies, or intravenously administered materials
* History of allergic/anaphylactoid-like reactions attributed to iodinated contrast agents or other components of the formulation
* Disturbances in normal fat metabolism, or total cholesterol greater than 240 mg/dL
* Pregnant or nursing women
* Exposure to significant radiation within 1 year, or previous CT scan within 5 years prior to check-in

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Assessment of safety by clinical laboratory parameters, vital sign measurements, electrocardiograms, and adverse event monitoring | Baseline and up to and including 28 days post drug administration

SECONDARY OUTCOMES:
Maximum blood concentration (Cmax), half-life (t1/2), and ratio of free to encapsulated circulating iodixanol | Baseline and up to 28 days post drug administration
Radiographic density in ROIs by abdominal CT imaging | From 3-5 hours and up to 72 hours following NCTX administration

CONTACTS AND LOCATIONS:
Overall Officials: Philip T Leese, MD, Principal Investigator — Quintiles Phase 1 Services
Locations (1):
- Quintiles Phase 1 Services, Overland Park, Kansas, United States